CLINICAL TRIAL: NCT02965560
Title: A Study on Biomarkers Predicting the Outcome of Acute-on-chronic Liver Failure
Brief Title: Exploring Biomarkers Predicting the Outcome of Acute-on-chronic Liver Failure
Acronym: PGE2
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Haihong Zhu, Professor, First Affiliated Hospital of Zhejiang University
Other Study IDs: tclouds
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2016-10

CONDITIONS: Acute-On-Chronic Liver Failure; Cirrhosis and Chronic Liver Disease
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- HC,CHB,AD,ACLF: HC healthy controls; CHB chronic hepatitis B; AD acute decompensated cirrhosis; ACLF acute-on-chronic liver failure.
  Interventions: Diagnostic Test: plasma suPAR, PGE2 measurement. Other biomarkers were just recorded from clinical laboratory.

INTERVENTIONS:
Diagnostic Test: plasma suPAR, PGE2 measurement. Other biomarkers were just recorded from clinical laboratory.

SUMMARY:
Acute-on-chronic liver failure (ACLF) is an ailment with high incidence of multiorgan failure (MOF) and consequent mortality. Systemic inflammation and susceptibility to infection are characteristic pathophysiological features. Prostaglandin E2 (PGE2) could subdue systemic inflammation and alleviate liver injury in mice model. However, there are no studies evaluating PGE2 as a predictor of early mortality.This study is designed to investigate whether plasma PGE2 and its receptors are associated with development of MOF and predict short-term mortality in patients with acute-on-chronic liver failure. By the way, we will also measure several other potential predictive factors (C-reactive protein,severe hyponatremia, Second infections,Diabetes mellitus,High density lipoprotein,interleukin-10,serum bile acids,ferritin,the neutrophil to lymphocyte ratio,soluable urokinase plasminogen activator receptor,vWF-Ag levels and FVIII-to-PC ratios).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute-on-chronic liver failure according to Asian-Pacific Association for the Study of the Liver (APASL) diagnostic criteria

Exclusion Criteria:

* Hepatocellular carcinoma(HCC)
* Portal vein thrombosis
* Pregnancy
* Human immunodeficiency virus (HIV)
* Patients who had received immunomodulator,or cytotoxic/immunosuppressive therapy within at least the preceding 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohorts will be selected from Provincial General Hospital
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 90 days
incidence of multiorgan failure | 90 days
all cause mortality | 30 days

REFERENCES:
- [Derived] Wang Y, Wu F, Chen C, Xu L, Lin W, Huang C, Yang Y, Wu S, Qi J, Cao H, Li G, Hong M, Zhu H. Soluble urokinase plasminogen activator receptor is associated with short-term mortality and enhanced reactive oxygen species production in acute-on-chronic liver failure. BMC Gastroenterol. 2021 Nov 17;21(1):429. doi: 10.1186/s12876-021-02006-x. PMID 34789156